CLINICAL TRIAL: NCT01417884
Title: Development of a Prospective Cardiovascular Patient Cohort and Biobank and Provision of Genomic Analyses With Focus on Platelet Function and Platelet Mediated Inflammatory Processes
Brief Title: Monocentric Registry to Investigate the Role of Platelet Function, Platelet Genetics, Proteomics and Metabonomics in Heart Disease
Acronym: TuePIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: National Heart and Lung Institute (Other); Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Prof. Dr. Tobias Geisler, Deputy Director, University Hospital Tuebingen
Other Study IDs: TuePIC012011; KFO 274/1-1 (Other Grant/Funding Number: German Research Council)
Record Dates: First submitted 2011-08-12; First posted 2011-08-16 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Cardiovascular Disease
Keywords: molecular cardiology; molecular epidemiology; platelets; cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, salivatory
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ischemic heart disease: stable coronary artery disease, acute coronary syndromes
- non-ischemic heart disease: inflammatory heart disease, heart failure (non-ischemic), valvular heart disease

SUMMARY:
Molecular targets on platelets are pivotal for the development of new pharmacological substrates for platelet inhibition and to better understand the impact of platelet-mediated inflammatory processes for the progression of heart disease, such as coronary heart disease and chronic heart failure. Previous investigations on the thienopyridine Clopidogrel have underlined the importance of combined risk factor analysis. Thus, clopidogrel´s prognostic efficacy relies on the combination of genetic factors (mainly polymorphisms of CYP2C19 encoding genes) and non-genetic factors, such as age, diabetes mellitus or concomitant drugs. Therefore, a prospective patient cohort with exact phenotypic characterisation according to standardized protocols is necessary to enable the examination of the clinical relevance of potential molecular targets. A supplementary provision of high quality bio-material enables the systematic examination of new promising platelet-biomarkers in cardiovascular disease, which already have produced significant results on experimental animal and/or cell biologic models. Primary objective of the central project is to establish a prospective cardiological cohort in the setting of a Cardiovascular Clinical Research Unit (CCRU) with an affiliated Biobank and thus to review the clinical significance of potential targets deriving from individual subprojects within the research group (German Research Council KFO 274/1-1) to safeguard a translational approach.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ischemic and non-ischemic heart disease
2. informed consent by patients or relatives in case of missing capacity to consent due to health status

Exclusion Criteria:

1. Patients <18 years
2. missing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In-hospital patients and outpatients
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2012-01; Primary Completion 2020-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 4 years

SECONDARY OUTCOMES:
Cardiovascular Death | 4 years
Myocardial infarction | 4 years
ischemic stroke | 4 years
bleeding | 4 years
stent thrombosis | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Geisler, Prof. Dr., Principal Investigator — UKT; Matthias Schwab, Prof. Dr., Principal Investigator — UKT, IKP Stuttgart
Locations (1):
- Medizinische Klinik und Poliklinik Tübingen, Cardiology Department, University Hospital Tübingen, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Borst O, Munzer P, Alnaggar N, Geue S, Tegtmeyer R, Rath D, Droppa M, Seizer P, Heitmeier S, Heemskerk JWM, Jennings LK, Storey RF, Angiolillo DJ, Rocca B, Spronk H, Ten Cate H, Gawaz M, Geisler T. Inhibitory mechanisms of very low-dose rivaroxaban in non-ST-elevation myocardial infarction. Blood Adv. 2018 Mar 27;2(6):715-730. doi: 10.1182/bloodadvances.2017013573. PMID 29588304